CLINICAL TRIAL: NCT02395913
Title: Compare Safety and Pharmacokinetic Properties of Surfolase Capsule(Acebrophylline 100mg) and Surfolase CR(200mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HT-002-02
Record Dates: First submitted 2015-02-10; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Male
MeSH Terms: interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- R (Active Comparator)
  Interventions: Drug: Surfolase capsule (100mg)
- T1 (Experimental)
  Interventions: Drug: Surfolase CR (200mg, T1)
- T3 (Experimental)
  Interventions: Drug: Surfolase CR (200mg, T3)
- T4 (Experimental)
  Interventions: Drug: Surfolase CR (200mg, T4)

INTERVENTIONS:
Drug: Surfolase capsule (100mg) — Surfolase capsule one capsule twice one days fasting administration
  Arms: R
Drug: Surfolase CR (200mg, T1) — one tablet once one days fasting administration.
  Arms: T1
Drug: Surfolase CR (200mg, T3) — one tablet once one days fasting administration.
  Arms: T3
Drug: Surfolase CR (200mg, T4) — one tablet once one days fasting administration.
  Arms: T4

SUMMARY:
Acebrophylline is metabolized by being separated into Ambroxol and 7-theophylline when orally administered as a salt composed of an acid-base as a compound that was synthesized by and chloride (salifying) the ambroxol to 7-theophylline. Acebrophylline is selectively applied to the bronchial or lung tissue and inhibit the activity of phospholipase bronchoalveolar shows the expectorant action to raise the surface activity of the alveolar, leukotrienes (LTs) and by suppressing the production of prostaglandins (PGs), showed potent anti-inflammatory activity, bronchial was celebrated by reducing the bronchial hyperreactivity to normal state is allowed to recuperate or extended.

It was developed to improve compliance improve pharmaceutically Surfolase capsule(Acebrophylline 100mg) that intake twice daily 100mg to Surfolase CR(Acebrophylline 200mg) that intake once daily 200mg

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 20 and 55 years, BMI >18.5, <25, inclusive

   *Body mass index (kg/m2) = weight(kg)/height(m)2
2. Subject who don't have congenital or chronic diseases and have no abnormal medical examination results.
3. Subject is healthy (no clinically relevant findings in any of the investigations of the pre-examination) as judged by the investigator
4. Subjects who signed and dated in informed consent form indicating that the subject has decided to participate in the study after being informed of all pertinent aspects of the study

Exclusion Criteria:

1. Subject with known for hypersensitivity reaction to acebrophylline, xanthine and food.
2. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
3. Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
4. Subject with known for history of gastrointestinal disease or gastrointestinal surgery which affect on the absorption drug
5. Subjects with any of the following condition in screening (blood pressure, 12-lead ECG, blood, urinalysis, etc.)
6. Subject with any of the following conditions in laboratory test i. AST(sGOT) or ALT(sGPT) > Upper normal limit × 1.25 ii. Total bilirubin > Upper normal limit × 1.5
7. If the estimated GFR < 80mL/min/1.76m2 using MDRD formula.
8. Systolic blood pressure <=90mmHg or diastolic blood pressure >=150mmHg or a person showing the corresponding figures <=50mmHg or >=100mmHg in vital signs.
9. Who has history of drug abuse (especially hypnotic, central acting analgesics, psychotropic drugs, such as opiates or central nervous system acting drug) or shows positive reactions to drug of abuse in urine drug screening tests.
10. Excessive caffeine and alcohol intake, smoking person(caffeine: > 5cups/day, alcohol: >210g/week, tobacco: > 10 cagarettes/day)
11. Use of any prescription medication within 14 days prior to study medication dosing or use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
12. Participation in any clinical investigation within 60days prior to study medication dosing
13. Subjects with whole blood donation within 60days, component blood donation within 30days
14. Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
AUCt of ambroxol | blood serum sampling
Cmax of ambroxol | blood serum sampling

SECONDARY OUTCOMES:
AUCinf of ambroxol | blood serum sampling
Tmax of ambroxol | blood serum sampling
t1/2 of ambroxol | blood serum sampling

CONTACTS AND LOCATIONS:
Overall Officials: Park, Principal Investigator — Yonsei University Health System, Severance Hospital